CLINICAL TRIAL: NCT03277495
Title: Predictors and Consequences of Combustible Cigarette Smokers' Switch to Standardized Research E-Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); University of Chicago (Other)
Responsible Party: Principal Investigator, Robin Mermelstein, Distinguished Professor and Director, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0948; 1U01DA045524-01 (NIH)
Record Dates: First submitted 2017-09-07; First posted 2017-09-11 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Participants will be stratified by sex and randomly assigned with a 1:1 allocation ratio to one of two conditions: 1) to receive SREC pods in their usual flavor (N = 60); and 2) to receive SREC pods in their choice of flavor (N = 60).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual SREC pods Flavor (Active Comparator): The liquid in the e-cigarette refills contains nicotine and comes in the following flavors: tobacco, menthol, blueberry, and watermelon. The participant will receive SREC pods in their usual flavor.
  Interventions: Behavioral: Brief behavioral counseling
- Choice of SREC pods Flavors (Active Comparator): The liquid in the e-cigarette refills contains nicotine and comes in the following flavors: tobacco, menthol, blueberry, and watermelon. The participant will receive SREC pods in their choice of flavor.
  Interventions: Behavioral: Brief behavioral counseling

INTERVENTIONS:
Behavioral: Brief behavioral counseling — Staff will engage in behavioral counseling to identify strategies for reducing combustible cigarette use. All participants in the trial receive this intervention

SUMMARY:
The primary goal of this study is to examine whether cigarette smokers can reduce their use of conventional, combustible cigarettes by switching to a Standardized Research E-Cigarette (SREC); whether participants can maintain these reductions and use of SRECs over a 12-week period; and whether there are changes in subjective and objective measures of health, appeal and acceptability of the products used during this time frame.

DETAILED DESCRIPTION:
The investigators will enroll 120 conventional cigarette smokers who report smoking at least 3 cigarettes/day. Following completion of baseline questionnaires and a week of ecological momentary assessments (EMA) tracking participants usual smoking behavior, participants will be stratified (by sex) and randomly assigned with a 1:1 allocation ratio to one of two conditions: 1) to receive SREC pods in their usual flavor (N = 60); and 2) to receive SREC pods in their choice of flavor (N = 60). The SREC pods used in this study come in tobacco, menthol, blueberry, and watermelon flavors. No other flavors will be available to use with the SREC.

Counseling at Week 2. Participants in both conditions will receive brief behavioral counseling on reducing their combustible cigarette use by substitution with SREC. Staff will work with participants to set individual goals for reduction during this first week, with the goal of achieving at least 75% reduction in the number of combustible cigarettes smoked by the end of the week, and all are encouraged to reduce further. Participants will also be told not to use any other combustible tobacco products. During the week, participants will complete a daily text or web report on number of cigarettes smoked and SREC pods used.

Week 3 Visit. Participants will bring back all used and unused pods for adherence counts, complete a brief questionnaire about subjective reactions and potential adverse effects, and provide breath CO. Participants will meet with study staff to review their progress with switching to SREC and receive continued behavioral counseling to substitute SREC for cigarettes. Participants will receive SREC refill pods and will start a second 7-day EMA protocol.

Week 4 Visit. EMA debriefing to check for compliance and any problem reports; return of used and unused pods, complete assessments; review of progress with switching to SREC. Participants will receive a 2 week supply of SREC pods.

Weeks 5-13. Participants return to the study office every 2 weeks to return pods, receive a new supply, and provide breath CO. During the week, participants will continue daily use reports via web/text.

Week 14 (End-of-Treatment). Participants return to the study office to complete a full assessment battery. They will be encouraged to continue to stay off/reduce all combustible cigarettes, but will not receive additional SREC refills from the study.

Week 18 (One Month Follow-up). Participants complete a final survey.

ELIGIBILITY:
Inclusion Criteria:

1. men and women 21 years of age or older;
2. daily smoking rate of 3 cigarettes/day or greater for at least one year;
3. interested in reducing cigarette use;
4. willing to try e-cigarettes;
5. able to attend in-person assessments over the next 5 months;
6. English speaking; and
7. breath CO of 3ppm or greater (assessed at baseline visit). Women who are of child-bearing age cannot be pregnant and must agree to use an approved form of birth control during the study.

Exclusion Criteria:

1. current use of any smoking cessation medication or participation in a smoking cessation program or study;
2. current daily ENDS user;
3. pregnancy if female; and
4. no two members of the same household may participate in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2024-08-14 (Actual); Study Completion 2024-08-14 (Actual)

PRIMARY OUTCOMES:
Combustible cigarette use | 12-weeks (end of treatment)
  number of cigarettes smoked per week

SECONDARY OUTCOMES:
Abstinence | 12-weeks (end of treatment)
  The proportion of participants who achieve total abstinence from combustible cigarettes (defined as no cigarette smoking in the past 7 days)
Number of cigarettes smoked | 18-weeks (end of trial)
  The total number of cigarettes smoked in the 7 days prior to the last assessment

OTHER OUTCOMES:
CO level | 12-weeks
  in ppm
Blood Pressure | 12-weeks
  systolic blood pressure and diastolic blood pressure in mm hg
Heart Rate | 12-weeks
  beats per minute
Weight | 12-weeks
  in pounds
self-report of respiratory symptoms | 12-weeks
  The St. George's Respiratory Questionnaire (SGRQ)
nicotine dependence | 12-weeks
  Fagerstrom Test for Nicotine Dependence

CONTACTS AND LOCATIONS:
Overall Officials: Robin Mermelstein, PhD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Institute for Health Research and Policy, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Within two years after the final data collection is completed, the investigators will create a completely de-identified data set will that obfuscate any variable that might potentially be used to identify an individual study participant. Data collection instruments, codebooks, and other data documentation will be made available in conjunction with this dataset in a standard format that is readable across a variety of applications and operating system platforms.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will become available no later than two years after the final data collection is completed. There is no time frame identified for stopping the sharing of the data.
Access Criteria: A data sharing agreement will be required for release of any data. Individuals requesting a copy of study data will need to submit a detailed research plan that includes the purpose of the proposed research, the variables required, the duration of the analysis phase, IRB approval with FWA information, investigator training in human subjects and other approvals specific to the individual datasets. They will also be required to submit a Data Protection Plan or Institutional Privacy Policy, describing the computing environment in which data will be managed and analyzed and how physical access to computing equipment will be controlled. Data will only be released once all IRB approvals and Human Subjects concerns have been addressed.